CLINICAL TRIAL: NCT03205007
Title: Adaptation of a Health Promotion Nutrition Program for Older Adults Entitled:Beneficial Bites for Healthy Living
Brief Title: Adaptation of a Health Promotion Nutrition Program for Older Adults
Acronym: BBHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 133-AAB8352; 2017-0188 (Other: IRB ID); A540300 (Other: UW Madison); NUR\FACILITIES OPRTN (Other: UW Madison)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-01

CONDITIONS: Nutrition Disorders in Old Age
Keywords: Health Promotion; Nutrition; Older Adults

STUDY DESIGN:
Intervention Model Description: Pre-Post changes in dietary behavior
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health promotion nutrition program (Experimental): Health promotion nutrition program
  Interventions: Behavioral: Health promotion nutrition program

INTERVENTIONS:
Behavioral: Health promotion nutrition program — Health promotion nutrition program

SUMMARY:
Our overarching goal is to prove the benefit of a behavior change intervention designed to help older people overcome barriers associated with risk for inadequate nutrition, so that they can improve their nutritional intake of fruits and vegetables, low fat dairy, whole grains, nuts, lean meats, poultry and fish.

DETAILED DESCRIPTION:
Our overarching goal is to prove the benefit of a behavior change intervention designed to help older people overcome barriers associated with risk for inadequate nutrition, so that they can improve their nutritional intake of fruits and vegetables, low fat dairy, whole grains, nuts, lean meats, poultry and fish. In this proposal, as a first step, we will build on the Beneficial Bites health promotion nutrition program (developed by Dietitians in northwestern Wisconsin), to produce "Beneficial Bites for a Healthy Life" (BBHL), which uses Social Cognitive Theory to change older adults' eating behaviors to minimize risks for inadequate nutrition for older adults. We will use a pre-post design to evaluate changes in dietary behavior 1 week and 6 months after the BBHL program. Our goal is to create a program that incorporates senior-specific nutrition information and recommendations as well as behavior change principles. There currently is no proven program that includes both of these components. This project is designed to provide data for a randomized trial for later testing so that it will eventually become eligible for future federal health promotion program funding (through Older Americans Act Title IIID funding) and thus be self-sustainable across Wisconsin and the rest of the nation.

Significance: Inadequate nutrition in older adults has been described as a crisis in America, which leads to increased illness and disability. This crisis is rapidly increasing as baby boomers age. A recent study looking at nutritional intake of older adults living in Pennsylvania found that 56% were at risk of inadequate nutrition2. Barriers to good nutrition include restricted finances leading to diets dominated by sugars, refined starches, and fatty meats; poor dental health, or problems chewing or swallowing food limiting healthy food choices; limited mobility making it difficult to shop for healthy foods; and lack of education on which foods are more nutrient dense leading to poor food choices. We propose to create a theory-based behavior change program that will not only provide nutrition education, but also will help older adults learn and incorporate into daily life strategies to minimize or overcome these common barriers to good nutrition. Current nutrition education programs tend to target a specific disease such as diabetes, heart disease, or osteoporosis, which may not be suitable for a general audience. Alternatively, a number of programs combine diet and exercise, but many older adults may be uninterested or unable to participate in exercise. Existing programs tend to focus more on providing education than on behavior change. Finally, no existing programs contain a maintenance component after the initial program is delivered.

Given the prevalence of inadequate nutrition, older adults should have access to proven nutrition behavior-change programs. The federal government recognizes this need, and through the Older Americans Act (OAA), provides funding to the states for programs that support healthy lifestyles and promote healthy behaviors. Beginning October 1, 2016, all health promotion programs using OAA Title IIID funds have to meet the following criteria: "Proven effective with an older adult population, using Experimental or Quasi-Experimental Design". Currently, there are no health promotion nutrition programs for older adults that meet these criteria. This creates a critical need for a behavior change nutrition program with proven effectiveness, which can be implemented in Wisconsin and nationally under OAA Title IIID funding.

Design and Aims:

Aim 1 To modify the BBHL program, based on Social Cognitive Theory to: 1) change older adults' eating behaviors to improve nutritional intake of fruits and vegetables, low fat dairy, whole grains, nuts, lean meats, poultry and fish, and 2) help older adults to successfully and sustainably utilize strategies to overcome barriers associated with risk of inadequate nutrition.

To address Aim 1, the Beneficial Bites program will be modified to produce a program entitled Beneficial Bites for a Healthy Life (BBHL). Overview of BBHL: This program will include 8 weekly 1.5 hour sessions designed to address common risks for inadequate nutrition faced by older adults, and help participants succeed in following a healthier diet building on behavior change techniques. The 8 sessions will promote fruits and vegetables, low or no fat dairy, whole grains, healthy fats, legumes and nuts, and lean meats, fish, and poultry. Each session will include: 1) group discussions with brain-storming to identify barriers and strategies to overcome barriers to eating a healthy diet; 2) an activity such as tasting different foods or playing nutrition related games; 3) homework, such as keeping a food diary (self-monitoring), or selecting nutritional foods when shopping (self-efficacy); and 4) feedback on performance of outside activities. When the 8 week program ends, a 6 month home program will begin. The dietitian will continue to monitor the participants with monthly coaching telephone calls designed to enhance maintenance of BBHL behavior change principles.

Dietitians from the Aging and Disability Resource Center of Barron, Rusk & Washburn Counties, Darby Simpson, Jennifer Jako, and Leslie Fijalkiewicz, will prepare content for the 8 sessions. They are experienced in delivering evidence based health promotion programing for older adults and understand their target audience. The investigators in Madison will develop theory-driven behavior change programing to integrate into the sessions. Co-investigator Kimberlee Gretebeck previously developed behavior change lessons incorporating Social Cognitive Theory for a proven program, Physical Activity for Seniors for Life (PALS), which is being disseminated through ADRCs in 8 counties in Wisconsin, in preparation for statewide dissemination. The behavior change techniques and strategies used successfully in PALS (goal setting, barrier identification/problem solving, self-monitoring, relapse prevention, etc.) will be modified to relate to following a healthy diet. The nutrition content will then be merged with the behavior change component. The merged sessions will then be sent back to the dietitians for review and comment. It is anticipated that 2-3 revisions will be needed. BBHL will then be offered with 10 participants at the Senior Center in Cameron Wisconsin. After participating in BBHL, we will conduct a focus group with participants and interviews with BBHL leaders to determine what content to keep or omit. Responses will be used to revise BBHL. BBHL will be revised prior to starting Aim 2.

Aim 2 Evaluate the modified BBHL for effectiveness of change in nutrient intake and nutrition behavior by subjective and objective measurement 1 week and 6 months after program completion. We hypothesize that participants will show improvements in the intake of fruits and vegetables, low or no fat dairy, whole grains, healthy fats, legumes and nuts, and lean meats, fish, and poultry one week and 6 months after the program compared to baseline (before beginning BBHL).

To address Aim 2, BBHL will be offered once at the Cumberland Senior Center and twice at the Rice Lake Senior Center. A total of 30 participants (10 per group times 3 groups) will be recruited by the dietitians and support staff from the ADRC of Barron, Rusk & Washburn Counties using the recruiting methods they use for other evidence based health promotion programs they provide. Eligibility criteria to participate includes no severe dietary restrictions (kidney disease), and the ability to make independent food choices and prepare meals (individuals being provided with meals will be excluded). Moderate dietary restrictions associated with chronic diseases such as diabetes can be accommodated within the program. Before BBHL begins, after completing the 8 sessions, and after completing the 6 month maintenance period with coaching phone calls, participants will complete validated standardized questionnaires on food intake and nutrition behavior.

The knowledge we gain from this pilot work will benefit not only the ADRC of Barron, Rusk, and Washburn counties with whom we are collaborating but the entire Aging Network of Wisconsin. If this program is shown to be beneficial based on pre-post data, then we will apply for Federal funding to conduct a randomized, controlled trial to prove effectiveness. Ultimately, we hope to create a proven program to improve nutritional intake by older adults. Once proven, we will work with Wisconsin's Aging Network and the Wisconsin Institute for Healthy Aging, to disseminate the program across the state of Wisconsin and nationally.

ELIGIBILITY:
Inclusion Criteria:

Independent

Exclusion Criteria:

Kidney Disease -

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Dietary Behavior | 8 weeks
  Block FFQ, Metabolomics

SECONDARY OUTCOMES:
Dietary Behavior | 6 Months
  Block FFQ, Metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Randall Gretebeck, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin-Madison, Madison, Wisconsin
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No